CLINICAL TRIAL: NCT05819294
Title: A Feasibility Study of the Diagnostic Yield of Pre-aspiration Pleural Fluid Agitation in Non-infected Pleural Effusion
Brief Title: Diagnostic Yield of Agitated Exudative Non-infected Pleural Effusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Salama Sadaka, Lecturer, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0305913
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Pleural Effusion
Keywords: pleural effusion; exudate
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Intervention Model Description: All participants will undergo both thoracentesis techniques; the standard and the experimental pre-aspiration agitated fluid techniques
Masking Description: Laboratory personnel responsible for the cytological and biochemical analysis will be blinded to the identity of the paired samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard thoracentesis followed by pre-aspiration fluid agitation (Experimental): Participants will undergo the standard thoracentesis followed by the experimental pre-aspiration fluid agitation technique
  Interventions: Procedure: Agitated Pleural Fluid Thoracentesis

INTERVENTIONS:
Procedure: Agitated Pleural Fluid Thoracentesis — Using a 16-18 gauge cannula, a standard thoracentesis will be performed then a sample of pleural fluid will be aspirated and rapidly flushed into the pleural space and redrawn again for a few cycles before a sample is finally drawn into the collection syringe

SUMMARY:
The goal of this study is to compare the diagnostic yield in terms of cellular content and biochemical characteristics of pre-aspiration agitated pleural fluid versus that of conventionally aspirated fluid in pleural infection patients. The hypothesis is that the agitated fluid would be more representative and thus may aid the diagnosis of non-infected exudative pleural effusions.

DETAILED DESCRIPTION:
Transudation or exudation are the two mechanisms by which fluid accumulates, where Starling forces' imbalance is responsible for the former and inflammatory increase in capillary permeability accounts for the latter. Despite the history and presentation commonly suggesting the underlying etiology, pleural fluid aspiration and analysis is frequently required for confirmation of the nature and cause of the effusion. Aspirated pleural fluid is routinely subjected to biochemical analysis as well as microbiological and cytological analysis especially when infection or neoplasia is suspected. One drawback however to thoracentesis analysis is the relatively low diagnostic yield in different forms of exudative effusion. Tuberculous pleural effusions have a yield of <10% on acid-fast bacilli smears and overall yield <30% on solid culture. Conventional cytologic analysis from malignant pleural effusions also show a relatively low overall yield of around 51%, though this could be highly variable depending on the primary cancer involved (6% in mesothelioma - 80% in ovarian adenocarcinoma).In addition, it is not uncommon for analysis results to widely vary in the same patient in those with loculated and in malignant pleural effusions. This could be attributed to the compartmentalization in complex septated collections and heterogenous distribution of cellular components throughout the pleural space. The gold standard however in diagnosing unexplained exudative pleural effusions is pleural biopsy which is technically demanding and sometimes associated with longer hospital stay along with the increased incurred costs.

The investigators propose a method for improving the representativeness of pleural fluid samples via pleural agitation prior to aspiration in exudative noninfected pleural effusion. The aim is to test the feasibility and safety of using pleural fluid agitation prior to aspiration and to investigate the potential for an improved diagnostic yield using this novel thoracentesis technique in patients with exudative non-infected pleural effusion. A control group of 10 participants with transudative pleural effusion (based on history, clinical picture, and imaging) will be included to exclude any effect of the agitation procedure on the biochemical profile of the pleural fluid. These will include patients with uncontrolled heart failure, renal or hepatic impairment presenting with classical uncomplicated free pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. At least a moderate amount of pleural fluid collection (2 or more intercostal spaces on thoracic ultrasound)

Exclusion Criteria:

1. Minimal - mild pleural fluid deemed unsuitable for aspiration and agitation
2. Hemodynamic instability
3. Pleural infection based on clinical presentation, imaging or laboratory investigations and pleural fluid examination showing glucose < 40 mg/dL or pH <7.2 with lower respiratory infection, positive gram stain or bacterial culture or pus on aspiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of the cytological analysis | 14 days
  Percentage of samples with a positive cytological result among both aspiration techniques
Diagnostic yield of the microbiolocal analysis (mycobacterial / fungal) | 14 days
  Percentage of samples with a evidence of mycobacterial / fungal elements among both aspiration techniques
Incidence of adverse events with pre-aspiration fluid agitation | 14 days
  Percentage of patients with incidence of adverse events during or right after pre-aspiration fluid agitation including pneumothorax or significant pain or cough or oxygen desaturation

SECONDARY OUTCOMES:
Protein level difference between both aspiration method | results within 1 day of sampling
  Difference in Protein levels in the aspirated fluid via both techniques
Lactate dehydrogenase (LDH) level difference between both aspiration method | results within 1 day of sampling
  Difference in LDH levels in the aspirated fluid via both techniques
Glusose level difference between both aspiration method | results within 1 day of sampling
  Difference in glucose levels in the aspirated fluid via both techniques
Neutrophilic count difference between both aspiration method | results within 1 day of sampling
  Difference in neutrophilic count in the aspirated fluid via both techniques
Lymphocytic count difference between both aspiration method | results within 1 day of sampling
  Difference in lymphocytic count in the aspirated fluid via both techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Diseases Department, Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No